CLINICAL TRIAL: NCT00287287
Title: Phase II Trial of REVLIMID® (Lenalidomide) for Therapy of Radioiodine-Unresponsive Papillary & Follicular Thyroid Carcinomas
Brief Title: REVLIMID® (Lenalidomide) for Therapy of Radioiodine-Unresponsive Papillary and Follicular Thyroid Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Ain (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Kenneth Ain, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-701-F3R; NCT00381498 (obsolete NCT alias)
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Thyroid Neoplasms
Keywords: Lenalidomide; Clinical Trials phase II; Carcinomas, thyroid; Radioiodine-Unresponsive; Papillary; Follicular
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Revlimid) (Experimental): Treatment will be initated at 25 mg/day taken in the morning. Dose adjustments may be made to alleviate toxicities.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Initial dose is 25 mg/day dose will be adjusted accordingly as needed. Dose range for the study is 5 to 25 mg/day
  Other Names: Revlimid

SUMMARY:
The primary objective of the study is to assess the anti-tumor activity of REVLIMID® (lenalidomide), administered as a single agent, in patients with distantly metastatic thyroid carcinomas which are unresponsive to systemic radioiodine, in terms of tumor response and response duration.

DETAILED DESCRIPTION:
Thalidomide has found new uses as a tumor anti-angiogenesis agent that is capable of diminishing the proliferation of angiogenesis-dependent solid malignancies. Distantly metastatic, unresectable medullary thyroid carcinomas, as well as de-differentiated papillary and follicular thyroid carcinomas, which no longer concentrate radioiodine, have no known effective systemic therapies. We have verified, in the context of a completed phase 2 clinical trial, that thalidomide has significant activity in thyroid carcinomas that are no longer radioiodine avid and are rapidly progressive. This activity has only limited durability of around 7 months and is associated with significant toxicities of sedation, constipation and neuropathy.

REVLIMID® (lenalidomide) is an analog of thalidomide with the chemical name, alpha-(3-aminophthalimido) glutarimide. REVLIMID® is noted to be more potent than thalidomide in inhibiting the production of TNF-alpha. It has more than doubled the inhibition of microvessel growth at the same concentration as thalidomide in a rat aorta angiogenesis model as well as greatly enhanced activity as an IMiD. Most importantly, it lacks much of the toxicity of thalidomide, particularly in regards to somnolence, neuropathy, or biochemical effects. In fact, patients with multiple myeloma, known to be resistant to thalidomide, were still seen to exhibit clinical responses to REVLIMID®. This makes REVLIMID® an appropriate agent to investigate in a phase 2 trial in thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of follicular, papillary, insular, or Hürthle-cell thyroid carcinoma. Histologic slides and/or tissue blocks must be reviewed at the University of Kentucky Medical Center.
* Patients must have an unresectable, distantly metastatic tumor, which does not concentrate radioactive iodine. Alternatively, follicular or papillary thyroid carcinoma patients with large distant tumor burdens which have not sufficiently responded to more than 800 mCi I-131 cumulative therapy and are progressive (criteria #4) may be appropriate for inclusion.
* No systemic chemotherapy agents within 4 weeks of initiation of therapy.
* Patients must have 3 consecutive radiographic evaluations demonstrating a cumulative 30% increase in tumor volume over a period of one year or less.
* Patients must be over the age of 18 years with the ability to understand and willing to sign an informed consent.
* Non-pregnant (if female). Women of childbearing potential (fertile females) must have a negative serum or urine pregnancy test within one day of starting study drug. In addition, sexually active fertile female subjects must agree to adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation, intrauterine device, barrier contraceptive with spermicide; or vasectomized partner) while on study drug. Men must agree to use latex condoms when having sex with fertile women.
* Karnofsky performance status ≥ 70.
* Baseline laboratory studies:

  * absolute neutrophil count (ANC) > 1000/mm3
  * platelet count ≥ 100 K/mm3
  * creatinine ≤ 1.5 mg/dL, and
  * transaminase levels (AST/SGOT, ALT/SGPT) ≤ 2 x upper limit of normal (ULN) (or ≤ 5 x I:M if hepatic metastases are present)
* Disease free of other prior malignancies for ≥ 5 years, with the exception of currently treated basal cell/squamous cell carcinoma of the skin or "in-situ" carcinoma of the cervix or breast.
* Thyroid stimulating hormone (TSH, thyrotropin) levels must be suppressed with sufficient levothyroxine to be kept beneath the normal range of the assay.

Exclusion Criteria:

* Patients may not have had prior REVLIMID® therapy.
* No serious concomitant medical or psychiatric illness that might interfere with informed consent or conduct of the study, including active infections that are not controlled with medication.
* Patients must not be pregnant or breastfeeding.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum, characterized by a desquamating rash, while taking thalidomide or similar drugs.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Concurrent use of other anti-cancer agents or treatments, with the exception of thyrotropin-suppression by levothyroxine.
* All subjects with central nervous system involvement, with the exception of those subjects whose central nervous system metastases have been treated with either radiotherapy and/or surgery and remain asymptomatic with no evidence of active central nervous system disease (verified by computed tomography [CT] scan or magnetic resonance imaging [MRI]) for at least 6 months.
* Known to be positive for HIV or infectious hepatitis, type A, B, or C.
* Patients with medullary or anaplastic thyroid carcinomas are excluded. Patients whose disease is limited to bone metastases are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2010-07-06 (Actual); Study Completion 2010-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B Ain, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide (Revlimid)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide (Revlimid)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of patients who responded to treatment (either stable disease or complete response) based on total tumor volume measurements from CT scans.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide (Revlimid)
Number analyzed (Participants) | 25
Participants | 17

ADVERSE EVENTS:
Time Frame: 4 years
Description: Serious adverse events were defined as Grade 3 or higher.
Arm/Group | Lenalidomide (Revlimid)
All-Cause Mortality (participants affected / at risk) | 25/25
Serious Adverse Events (participants affected / at risk) | 25/25
Other Adverse Events (participants affected / at risk) | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Revlimid) (N=25)
Neutropenia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1
Rash (Social circumstances) | 1
Pulmonary Embolism (Vascular disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Revlimid) (N=25)
Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Weight Loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-09-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT00287287/Prot_SAP_000.pdf